CLINICAL TRIAL: NCT02662478
Title: Accuracy and Feasibility of a Morpho-anatomical Classification Oriented Laparoscopic Resection of Gastric Stromal Tumors in Advanced Laparoscopic Surgery Center: a Prospective Cohort Study
Brief Title: Laparoscopic Resection of Large Gastric Stromal Tumors
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Bahçeşehir University (Other); Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, General Surgery, Medical Park Gaziantep Hospital
Other Study IDs: MK-006-ST
Record Dates: First submitted 2016-01-18; First posted 2016-01-25 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Laparoscopic gastric resection; gastrointestinal stromal tumor; laparoscopic surgery
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — gastric resection material
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- primary gastric GIST: Consisted of all consecutive cases of primary gastric stromal tumors (PGST) that underwent laparoscopic surgery (LS).
  Interventions: Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Laparoscopic Surgery — Mid-point between the xiphoid and umbilicus was used to the entrance site of the telescope. Open trocar insertion was used in patients with history of open upper abdominal surgery; otherwise Veress needle established CO2 insufflations. The number, size and entry points of the other trocars were tailored according to the tumor location and size. In general, 2 to 4 additional trocars were used. All specimens were taken out of the abdomen through a suprapubic transverse incision in a sterile bag. Resection technique was determined by the size, number, location of the lesion, and surgical anatomy of the stomach. Lymph node dissection was not done as it is unnecessary.

SUMMARY:
Despite laparoscopic surgical treatment has not been recommended in patients with gastric gastrointestinal stromal tumors (GIST) larger than 5 centimeter, but it continues to evolve rapidly to overcome the boundaries. Therefore the authors generated a morpho-anatomical classification system (MACS) adapted for primary gastric GISTs, by which they could plan to tailor the laparoscopic gastric resection appropriately. The aims of the study was to demonstrate the feasibility of laparoscopic surgery for primary gastric GISTs larger than 5 cm, to find out the accuracy and practicality of the MACS for the development a preoperative strategy and the extent to which this strategy overlaps with the reality.

DETAILED DESCRIPTION:
Incidence rate of gastrointestinal stromal tumors (GIST) is 10-15 per million per year. Although very rare, it is the most common mesenchymal tumor of the gastrointestinal tract, and the stomach is the most common affected organ with up to 55.6%. Despite recent drug discoveries have greatly impacted the treatment, complete surgical resection with adequate safety margin is still the only potentially curative treatment for primary gastric GIST with no evidence of metastasis. As sarcomas in general, most GISTs also metastasize hematogenously to the liver, disseminate peritoneally, and rarely show lymph node metastasis, therefore systematic or prophylactic lymph node dissection is usually unnecessary; a pick-up sampling is considered sufficient when a perilesional lymph node enlargement is found. In addition to that, these tumors tend to be soft and friable. Therefore pseudocapsule may be tearing spontaneously or inadvertently during surgery and tumor cells can be disseminating intraperitoneally which results in increased risk for recurrence and decreased survival.

Considering these properties of the tumor, the goals of surgery for primary gastric GIST are handling the tumor with great care to avoid tumor rupture as well as performing a complete resection with a negative surgical margin and preserving the organ function as much as possible. This can be accomplished by the traditional open, or more recently by the various total or hybrid laparoscopic techniques. Despite laparoscopic surgical treatment of the GISTs had not been recommended owing to the higher risk of tumor rupture and subsequent peritoneal seeding in consensus meetings in the United States and Europe in 2004 and 2005 respectively, it has experienced a rapid and major evolutionary process and currently it is being advised to be a standard approach for gastric GISTs irrespective of its size or location.

In addition to achieve an R0 resection without a tear in the tumor, the most important issue for the laparoscopic gastric GIST surgery is the preserving the function and not to cause a stenosis in the stomach as much as possible. According to the morphologic characteristics of the tumor and the area in the three-dimensional anatomical configuration of the stomach that involved by the tumor, a lot of laparoscopic surgical scenarios can be produced. Among them, to achieve the best alternative which meets all above criteria the authors generated a morpho-anatomical classification system by which they could plan preoperatively to tailor the gastric resection and all operational requirements. This system was partly inspired by the TNM classification for GISTs and Japanese classification of gastric carcinoma, has long been used in authors' institution when planning a laparoscopic intervention for various gastric lesions in patients in whom an appropriate preoperative patient evaluation is needed. It is then specifically composed and standardized to adapt for primary gastric GISTs and it was being used for large tumors up to 10 cm.

The aims of the study was to demonstrate the feasibility of laparoscopic surgery for primary gastric GISTs larger than 5 cm, to find out the accuracy and practicality of the classification system in the development a preoperative strategy and the extent to which this strategy overlaps with the reality.

ELIGIBILITY:
Inclusion Criteria:

* All patients with gastric GIST underwent laparoscopic surgery

Exclusion Criteria:

* Patients with GIST of other than stomach
* Patients who refused laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Using the Turkish national procedural classification code number for laparoscopic stomach surgeries, a search was made in the Medical Park Gaziantep Hospital database which identified 124 patients underwent laparoscopic gastric resection for tumor. Then an additional similar search was performed to obtain primary gastric GIST subgroup according to the histopathological results and a total of 23 patients in whom LRS were performed, were identified.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Success rate | within the first 30 days after surgery
  Laparoscopic surgery performed without conversion to open surgery with a negative surgical margin

SECONDARY OUTCOMES:
Accuracy of classification system | within the first 3 months after completion of the patient recruitment
  the rate of overlapping preoperative strategy with the postoperative reality

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Study Director — Bahçeşehir Üniversitesi Tıp Fakültesi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soreide K, Sandvik OM, Soreide JA, Giljaca V, Jureckova A, Bulusu VR. Global epidemiology of gastrointestinal stromal tumours (GIST): A systematic review of population-based cohort studies. Cancer Epidemiol. 2016 Feb;40:39-46. doi: 10.1016/j.canep.2015.10.031. Epub 2015 Nov 24. PMID 26618334
- [Background] Joensuu H, Vehtari A, Riihimaki J, Nishida T, Steigen SE, Brabec P, Plank L, Nilsson B, Cirilli C, Braconi C, Bordoni A, Magnusson MK, Linke Z, Sufliarsky J, Federico M, Jonasson JG, Dei Tos AP, Rutkowski P. Risk of recurrence of gastrointestinal stromal tumour after surgery: an analysis of pooled population-based cohorts. Lancet Oncol. 2012 Mar;13(3):265-74. doi: 10.1016/S1470-2045(11)70299-6. Epub 2011 Dec 6. PMID 22153892
- [Background] Demetri GD, von Mehren M, Antonescu CR, DeMatteo RP, Ganjoo KN, Maki RG, Pisters PW, Raut CP, Riedel RF, Schuetze S, Sundar HM, Trent JC, Wayne JD. NCCN Task Force report: update on the management of patients with gastrointestinal stromal tumors. J Natl Compr Canc Netw. 2010 Apr;8 Suppl 2(0 2):S1-41; quiz S42-4. doi: 10.6004/jnccn.2010.0116. PMID 20457867
- [Background] Han D, Deneve J, Gonzalez RJ. Recurrence risk after resection of gastrointestinal stromal tumors: size is not all that matters... The consequences of tumor rupture. Am Surg. 2012 Jan;78(1):74-9. PMID 22273319